CLINICAL TRIAL: NCT05897970
Title: Association Between 4-Month Isokinetic Testing Measures and Second Knee Injuries After
Brief Title: Association Between 4-Month Isokinetic Testing Measures and Second Knee Injuries After Primary Anterior Cruciate Ligament Reconstruction
Acronym: PREDICT-ACLv2
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: PREDICT-ACLv2
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2023-06

CONDITIONS: ACL Injury; Knee Injuries; Muscle Weakness
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACLR patients with Return-to-sport (RTS) follow-up: All sports patients who had a muscle evaluation at 3-4 months after ACLR since January 2017
  Interventions: Diagnostic Test: Return-to-sport (RTS) follow-up

INTERVENTIONS:
Diagnostic Test: Return-to-sport (RTS) follow-up — All sports patients who had a muscle evaluation at 3-4 months after ACLR since January 2017

SUMMARY:
Anterior cruciate ligament (ACL) is a frequent and disabling injury in athletes. Most of the time, ACL reconstruction (ACLR) is consider for regaining function and returning to preinjury sports while reducing the risk of secondary injuries. However, the risk of secondary severe knee injury is increased after ACLR, especially in athletes returning to strenuous activities. If strength symmetry is considered as an important factor in the Return-to-sport (RTS) decision, there is conflicting data about the association between strength symmetry and the risk of second knee injury after ACLR. The main objective of this study was to test if knee muscles strength symmetry at 4 months was associated with the psychological readiness and incidence of subsequent severe injury of both knees at a minimum 2 years follow-up after ACL-R.

ELIGIBILITY:
Inclusion Criteria:

Patients who have had an ACL reconstruction surgery (isolated or associated with other meniscal or ligamentary surgery) Patient included in the sport medicine follow-up protocole with intermediate and final isokinetic muscular assessment at 3-4 months Patient who received the information form Patients with access to the Internet

Exclusion Criteria:

Patient who did not participate in all follow-up consultations and isokinetic muscular assessments Patients who had a previous knee surgery before the ACLR Cognitive or sensory impairment making it impossible to understand the information form Neurological, traumatic or osteoarticular history responsible for muscle imbalance prior to surgery

Ages: 16 Years to 55 Years | Sex: All
Age Groups: Child, Adult
Study Population: All sports patients included in the sport medicine follow-up protocole with isokinetic muscular assessment at 3-4 months after ACL reconstruction surgery since January 2017 with a minium 2 years follow-up in the sports medicine department, Return To Sport Process
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Strength | ACL group: Two evaluations on both injured and healthy knees: 3-4 months after surgery; Routine practice following guidelines]
  Measurement of knee extensors and flexors peak strength (in newton.meter, Nm) on isokinetic dynamometer.

SECONDARY OUTCOMES:
Individual characteristics | ACLR group: Two follow-up medical consultations: (1) 4 months after surgery and (2) 2 years after the surgery for return to sport and reinjury;
  Personal characteristics recorded in the medical report as age, gender, type of sport and sport level of practice and return to sport after the surgery and severe reinjury on the operated knee or contralateral knee.
Surgery characteristics | ACLR group: Two follow-up medical consultations 4 months after surgery
  Surgery characteristics recorded in the medical report as the type of surgery, the surgery duration
Re-injuries | ACLR group: One evaluation with a minimum 2 years follow-up after the surgery
  Web based questionnaire about any sever knee injury (meniscus or ACL) after the primary ACLR
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) scale. | ACLR group: One evaluation with a minimum 2 years follow-up after the surgery
  Web based questionnaire with completion of the Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided